CLINICAL TRIAL: NCT00915811
Title: Pilot Study of Reduced Intensity Haematopoietic Stem Cell Transplantation in Patients With Poor Risk Myelodysplastic Syndrome and Acute Myeloid Leukaemia Utilising Conditioning With Fludarabine, Busulphan and Thymoglobulin
Brief Title: Pilot Study of Reduced Intensity Haematopoietic Stem Cell Transplantation in Patients With Poor Risk Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukaemia (AML) Utilising Conditioning With Fludarabine, Busulphan and Thymoglobulin
Acronym: FB-ATG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FB ATG is now a standard for sib allo MDS patients
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Professor Ghulam Mufti, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06CC12; REC - 06/Q0703/208; EudraCT - 2006-004452-20
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-06

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute
Keywords: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Haematopoietic stem cell transplantation; Fludarabine; Busulphan; Thymoglobuline
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — fludarabine; Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FBATG (Experimental): Haematopoietic stem cell transplantation utilising conditioning with Fludarabine, Busulphan and Thymoglobuline
  Interventions: Drug: Fludarabine; Drug: Busulphan; Drug: Thymoglobuline (Anti-thymocyte globulin [rabbit]) - Genzyme; Procedure: Haematopoietic stem cell infusion

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30mg/m2 intravenously daily on days -9 to -5 inclusive of stem cell infusion.
Drug: Busulphan — Busulphan 0.8mg/kg intravenously 6 hourly on days -4 and -3 of stem cell infusion.
Drug: Thymoglobuline (Anti-thymocyte globulin [rabbit]) - Genzyme — Thymoglobuline will be given intravenously over a minimum of 6 hours for the first two doses and 4 hours for the subsequent doses. Acute side effects of ATG appear to be reduced if a very low dose is given for the first injection. Thymoglobuline 0.5mg/kg iv on day -4, 1.5mg/kg/day on day -3; and 2mg/kg/day iv on day -2 to -1 inclusive.
Procedure: Haematopoietic stem cell infusion — The source of stem cells will be PBSC wherever possible. Patients whose donors decline or are unable to donate PBSC will be transplanted with marrow cells.

SUMMARY:
The purpose of this study is to determine the safety and feasibility of conditioning with fludarabine, busulphan and thymoglobuline in patients with myelodysplastic syndrome (MDS), myelodysplastic/myeloproliferative disorders (MDS/MPD) or acute myeloid leukaemia (AML) undergoing haematopoietic stem cell allograft with granulocyte colony-stimulating factor (G-CSF)-mobilised peripheral blood stem cells (PBSC) (or bone marrow) from HLA compatible sibling donors.

ELIGIBILITY:
Inclusion Criteria:

Patient Selection

1. Availability of a HLA compatible sibling donor
2. Age >18 years
3. Myelodysplastic Syndromes with IPSS Intermediate-2 or High.
4. Poor risk acute myeloid leukaemia, de novo or transformed from MDS
5. Ineligibility for standard conditioning allograft due to age or co-existing morbidities

Donor selection

1. Related donors compatible for HLA-A, B, C, DRB1 and DQB1 by molecular typing.

Exclusion Criteria:

Patient selection

1. Cardiac insufficiency requiring treatment or symptomatic coronary artery disease.
2. Hepatic disease, with AST > 2 times normal.
3. Severe hypoxaemia, pO2 < 70 mm Hg, with decreased DLCO < 70% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 60% of predicted.
4. Impaired renal function (creatinine > 2 times upper limit of normal or creatinine clearance < 50% for age, gender, weight).
5. Patients who have received previous treatment with Thymoglobuline
6. HIV-positive patients.
7. Female patients who are pregnant or breast feeding due to risks to foetus from conditioning regimen and potential risks to nursing infants.
8. Life expectancy severely limited by diseases other than MDS or MPD.
9. Serious concurrent untreated infection
10. Patients with limited life expectancy for other reasons
11. Serious psychiatric/ psychological disorders
12. Absence of /inability to provide informed consent

Donor selection

1. Age >75 years, unless independently assessed to be medically fit to donate
2. Donors who for any reason are unable to tolerate the leukapheresis procedure and cannot undergo anaesthesia for marrow harvest.
3. Donors who are HIV-positive, or hepatitis B or C PCR positive.
4. Donors who are medically unsuitable to donate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Treatment related mortality to Day 100 | Days 28, 56 and 100

SECONDARY OUTCOMES:
Incidence of single or multi-organ acute toxicity | Days 28, 56 and 100
Incidence of graft failure/rejection | Days 28, 56 and 100
Incidence of acute graft-versus-host disease | Days 28, 56, 100 and months 6, 9, 12, 18 and 24
Incidence of systemic infections | Days 28, 56, 100 and months 6, 9, 12, 18 and 24
EBV activation | Fortnightly for first 6 weeks after transplantation and then weekly for the first 6 months.
Overall survival | Days 28, 56, 100 and months 6, 9, 12, 18 and 24
Disease free survival/relapse risk | Days 28, 56, 100 and months 6, 9, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam J Mufti, MB, DM, FRCP, FRCPath, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom